CLINICAL TRIAL: NCT04791540
Title: Observational Pilot Study in Patients Who Underwent Tracheostomy: Sarcopenia Assessment by Handgrip Strenght and BIA. Association to Malnutrion Risk, Nutritional Status, Gut Microbioma and Decannulation Time.
Brief Title: Sarcopenia and Nutritional Status in a Rehabilitation Setting
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Florence (Other)
Responsible Party: Sponsor
Other Study IDs: SARCOBIA1_FDG
Record Dates: First submitted 2021-02-22; First posted 2021-03-10 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia
Keywords: handgrip strenght; bioelectrical impedance analysis (BIA); respiratory rehabilitation; tracheostomy decannulation; gut microbiota; GLIM criteria; MUST
MeSH Terms: conditions — Sarcopenia | interventions — Gastrointestinal Microbiome; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with trachestomy: Patients, attending a respiratory rehabilitation program, who underwent tracheostomy decannulation
  Interventions: Diagnostic Test: handgrip strenght; Diagnostic Test: Bioelectrical Impedance Analysis (BIA); Diagnostic Test: MUST; Diagnostic Test: GLIM; Biological: Gut microbiota; Biological: Blood Sample; Other: Anthropometric measures

INTERVENTIONS:
Diagnostic Test: handgrip strenght — Muscle strenght measured with a handheld dynamometer, at admission (T0) and at decannulation time (T1)
Diagnostic Test: Bioelectrical Impedance Analysis (BIA) — Muscle mass evaluated by Bioelectrical Impedance Analysis (BIA), at admission (T0) and at decannulation time (T1)
Diagnostic Test: MUST — Malnutrition risk assessed by Malnutrition Universal Screening Tool (MUST), at admission (T0) and at decannulation time (T1)
Diagnostic Test: GLIM — Malnutrition diagnosis performed by Global Leadership Initiative on Malnutrition (GLIM) criteria, at admission (T0) and at decannulation time (T1)
Biological: Gut microbiota — A fecal sample obtained at admission (T0) and at decannulation time (T1)
Biological: Blood Sample — A Blood sample obtained at admission (T0) and at decannulation time (T1)
Other: Anthropometric measures — Measurement of weight and height (assessed only at admission) to calculate the Body Mass Index (BMI), at admission (T0) and at decannulation time (T1)

SUMMARY:
In this pilot observational study the primary outcome is to assess, in a Respiratory Rehabilitation Unit, if there is an association between sarcopenia, assessed by handgrip strenght and BIA, and a delayed decannulation time in patients who underwent tracheostomy.

Secondary outcomes are to assess if there is an association between an increased malnutrition risk (assessed by MUST), a poor nutritional status (assessed by GLIM criteria) and a delayed decannulation time and the gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from patients or legal guardians for patients unfit to plead
* Presence of tracheostomy at admission

Exclusion Criteria:

* Refusal
* Pregnancy
* Pace maker/implantable cardioverter
* No legal guardians for patients unfit to plead

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent tracheostomy before admission, attending a rehabilitation program
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from admission in muscle mass at decannulation time | Respiratory Rehabilitation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Measurement of muscle mass with Bioelectrical Impedance Analysis (BIA).
Change from admission in hangrip strenght at decannulation time | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Measurement of handgrip strenght with a handheld dynamometer. Male cut-off: <27 Kg Female cut-off: <16 Kg

SECONDARY OUTCOMES:
Change from admission in Body Mass Index (BMI) score at decannulation time | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Measurement of height and weight to get a BMI score (weight/(height^2). BMI <18.5 Kg/m^2: underweight BMI 18.5-24.9 Kg/m^2: normal range BMI 25.0-29.9 Kg/m^2: overweight BMI 30.0-34.9 Kg/m^2 obese class I BMI 35.0-39.9 Kg/m^2 obese class II BMI >= 40 Kg/m^2 obese class III
Change from admission in Malnutrition Universal Screening Tool (MUST) score at decannulation time | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  MUST is a screening tool to identify adults who are malnourished, at risk of malnutrition or obese.
  score 0: low risk score 1: medium risk score 2 or more: high risk
Change from admission in nutritional status at decannulation time | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Global Leadership Initiative on Malnutrition (GLIM) criteria are 5 diagnostic criteria to assess malnutrition that include 3 phenotypic (weight loss, low body mass index and reduced muscle mass) and 2 etiologic (reduced food intake/assimilation, and inflammation/disease burden) criteria.
  To diagnose malnutrition at least 1 phenotypic criterion and 1 etiologic criterion should be present.
Change from admission in Gut Microbiota (GM) composition at decannulation time | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Gut Microbiota (GM) composition
Protein C reactive (PCR) | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in Protein C reactive (PCR) at decannulation time
Lymphocyte count | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in lymphocyte count at decannulation time
Creatinine | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in creatinine at decannulation time
Creatine Poshokinase | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in creatine poshokinase at decannulation time
Total serum protein | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in total serum protein at decannulation time
Albumin | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in albumin at decannulation time
Vitamin (25OH) D | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in vitamin (25OH) D at decannulation time
Selenium | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in selenium at decannulation time
Leptin | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in leptin at decannulation time
Uric Acid | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in uric acid at decannulation time
Magnesium | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in magnesium at decannulation time
Growth Hormone (GH) | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in growth hormone at decannulation time
Insuline-like Growth Factor-1 (IGF-1) | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in Insuline-like Growth Factor-1 (IGF-1) at decannulation time
Dehydroepiandrosterone (DHEA) | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in dehydroepiandrosterone (DHEA) at decannulation time
Testosterone | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in testosterone at decannulation time
Pro-inflammatory cytokine interleukin IL-6 | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in pro-inflammatory cytokine interleukinIL-6 at decannulation time
Tumor Necrosis Factor-α (TNF-α) | Respiratory Rehabiliation Unit admission (T0) and decannulation time (T1), an average of 10 days
  Change from admission in Tumor Necrosis Factor-α (TNF-α) at decannulation time

CONTACTS AND LOCATIONS:
Overall Officials: Chiara F Gheri, MD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats AJS, Crivelli AN, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee, GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. J Cachexia Sarcopenia Muscle. 2019 Feb;10(1):207-217. doi: 10.1002/jcsm.12383. PMID 30920778
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Manuel Gomez J, Lilienthal Heitmann B, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, M W J Schols A, Pichard C; ESPEN. Bioelectrical impedance analysis-part II: utilization in clinical practice. Clin Nutr. 2004 Dec;23(6):1430-53. doi: 10.1016/j.clnu.2004.09.012. PMID 15556267
- [Background] Kutsukutsa J, Mashamba-Thompson TP, Saman Y. Tracheostomy decannulation methods and procedures in adults: a systematic scoping review protocol. Syst Rev. 2017 Dec 4;6(1):239. doi: 10.1186/s13643-017-0634-0. PMID 29202866
- [Background] Ticinesi A, Nouvenne A, Cerundolo N, Catania P, Prati B, Tana C, Meschi T. Gut Microbiota, Muscle Mass and Function in Aging: A Focus on Physical Frailty and Sarcopenia. Nutrients. 2019 Jul 17;11(7):1633. doi: 10.3390/nu11071633. PMID 31319564
- [Background] Toptas M, Yalcin M, Akkoc I, Demir E, Metin C, Savas Y, Kalyoncuoglu M, Can MM. The Relation between Sarcopenia and Mortality in Patients at Intensive Care Unit. Biomed Res Int. 2018 Feb 12;2018:5263208. doi: 10.1155/2018/5263208. eCollection 2018. PMID 29789798
- [Background] Prado CM, Purcell SA, Alish C, Pereira SL, Deutz NE, Heyland DK, Goodpaster BH, Tappenden KA, Heymsfield SB. Implications of low muscle mass across the continuum of care: a narrative review. Ann Med. 2018 Dec;50(8):675-693. doi: 10.1080/07853890.2018.1511918. Epub 2018 Sep 12. PMID 30169116